CLINICAL TRIAL: NCT01691989
Title: A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED,PHASE III STUDY TO ASSESS THE EFFICACY,SAFETY AND TOLERABILITY OF ALEGLITAZAR ADDED TO A SU OR ADDED TO A SU IN COMBINATION WITH MET IN PATIENTS WITH T2D INADEQUATELY CONTROLLED WITH SU MONOTHERAPY OR WITH SU + METFORMIN COMBINATION THERAPY
Brief Title: A Study of Aleglitazar in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Are Inadequately Controlled With Sulfonylurea Alone or Sulfonylurea Plus Metformin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WC28325
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- aleglitazar (Experimental)
  Interventions: Drug: aleglitazar
- placebo (Experimental)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aleglitazar — 150 mcg orally once a day for 26 weeks
  Arms: aleglitazar
Drug: placebo — oral doses once a day for 26 weeks
  Arms: placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will assess the efficacy, safety and tolerability of aleglitazar compared with placebo when added to a sulfonylurea monotherapy or sulfonylurea plus metformin combination therapy in patients with type 2 diabetes mellitus who are inadequately controlled with sulfonylurea alone or sulfonylurea plus metformin therapy. Patients will be randomized to receive oral doses of 150 mcg aleglitazar once daily or placebo. The anticipated time on study treatment is 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of diabetes mellitus, type 2
* Patients treated with stable sulfonylurea monotherapy or sulfonylurea plus metformin combination therapy for at least 12 weeks prior to screening
* HbA1c >/=7% and </=9.5% at screening or within 4 weeks prior to screening and at pre-randomization visit
* Fasting plasma glucose </=240 mg/dL at pre-randomization visit
* Agreement to maintain diet and exercise habits during the study

Exclusion Criteria:

* Patients with Type 1 diabetes mellitus, secondary diabetes, diabetes resulting from pancreatic injury, or acute metabolic diabetic complications within the past 6 months
* Any previous treatment with thiazolidinedione or a dual PPAR agonist
* Any body weight lowering or lipoprotein-modifying therapy within 12 weeks prior to screening (except stable dose of statin)
* Any anti-hyperglycemic medication other than sulfonylurea alone or in combination with metformin within 12 weeks prior to screening
* Symptomatic congestive heart failure classified as New York Heart Association class II-IV at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin HbA1c | From baseline to week 26

SECONDARY OUTCOMES:
Change in lipid profile | From baseline to week 26
Change from baseline in fasting plasma glucose | From baseline to week 26
Responder rate as defined of hemoglobin HbAc1 <7.0% (<6.5%) | From baseline to week 26
Change from baseline in homeostatic index of insulin sensitivity (HOMA-IS) | From baseline to week 26
Change from baseline in markers of insulin sensitivity and cardiovascular risk | From baseline to week 26
Safety: incidence of adverse events | 30 weeks (26 weeks treatment and 4 weeks follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (15):
  - Chino, California
  - Los Angeles, California
  - San Diego, California
  - Santa Ana, California
  - Jacksonville, Florida
  - Kissimmee, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Avon, Indiana
  - Bethesda, Maryland
  - Durham, North Carolina
  - Morrisville, Pennsylvania
  - Greer, South Carolina
  - Dallas, Texas
  - Richmond, Virginia
- Argentina (3):
  - Buenos Aires
  - Caba
  - Rosario
- Colombia (3):
  - Bogotá
  - Floridablanca
  - Medellin-Antioquia
- Guatemala City, Guatemala
- Mexico (4):
  - Aguascaliente
  - Celaya
  - Guadalajara
  - Querétaro

REFERENCES:
- [Derived] Henry RR, Buse JB, Wu H, Durrwell L, Mingrino R, Jaekel K, El Azzouzi B, Andjelkovic M, Herz M. Efficacy, safety and tolerability of aleglitazar in patients with type 2 diabetes: pooled findings from three randomized phase III trials. Diabetes Obes Metab. 2015 Jun;17(6):560-565. doi: 10.1111/dom.12455. Epub 2015 Apr 8. PMID 25728612